CLINICAL TRIAL: NCT05801081
Title: The Relationship Between Physical Activity Level and Reaction Time in University Students
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: reaction time
Record Dates: First submitted 2023-03-20; First posted 2023-04-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity
Keywords: reaction time
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active group: Participants will be divided into two groups according to their physical activity level using the International Physical Activity Scale. Individuals with high physical activity levels will be included in this group.
- Inactive Group: cipants will be divided into two groups according to their physical activity level using the International Physical Activity Scale. Individuals with low physical activity levels will be included in this group.

SUMMARY:
Reaction time, movement and total movement time are said to affect athletic performance.

The unit of time between giving a stimulus to the person and the beginning of the person's voluntary response to this stimulus is defined as the reaction time.

Recent studies have reported that reaction time may depend on gender differences, neuromuscular and neurophysiological factors, force production, structural and neural properties of muscles, and information processing speed.

DETAILED DESCRIPTION:
In recent studies, it has been reported that reaction time can be affected by parameters such as gender, neuromuscular and neurophysiological factors, force production, structural and neural properties of muscles, and information processing speed. Reaction time measurements are basically for two functions. The first of these is the situations that we encounter during traffic lights, sportive activities or daily life activities. The other is to measure the duration of mental activities such as processing the stimulus from the environment, making decisions, programming the reaction.

Physical activity is defined as all movements that require energy expenditure as a result of the use of skeletal muscles. Physical activity has positive effects on the development of muscle strength, balance, flexibility, posture, reaction time and motor skills. There is a complex relationship between physical activity and cognitive performance. Depending on the chosen cognitive task and the type of exercise, there is a change in cognitive load.

ELIGIBILITY:
Inclusion criteria;

* Being between the ages of 20 - 30,
* Healthy individuals,
* Absence of carpal tunnel syndrome, Exclusion criteria ;
* Not having a musculosketal or neurological disease that limits mobility
* Absence of upper extremity sequelae,

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The 'Phalen Test' will be applied in order to eliminate the risk of finding a carpal tunnel for the people included in the study. The subjects included in the study will be classified according to their physical activity status by giving the "International Physical Activity Questionnaire (Short)". Records of the subjects' dominant hands will be taken and included in the analysis process.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Nelson Hand Reaction Test | Day 1
  A ruler is used for the Nelson hand reaction test. Sit on the chair in a comfortable position with the forearm and hand on the table. Thumb and index finger tips are brought in parallel to each other 8-10 cm outside the table. The ruler is held between the thumb and forefinger. In this position, the test ruler is released and the ruler is asked to catch it. The value at the top of the thumb is saved when the ruler is captured. A total of five attempts are made and the best three results are averaged and noted.
Reaction Time Measurement with Computer | Day 1
  Reaction time is recorded through a program on computers or tablets. The alerts sent are in visual or auditory form. In reaction measurement, stimuli appear on the screen (5-15 seconds), which are not clear when. In order to eliminate the resulting image or auditory stimulus, it gives by pressing the specified key on the keyboard or screen. The applied test is recorded by the computer. A total of five attempts are made. It is noted by averaging the three best results.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire Short Form (IPAQ-SF) | Day 1
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klasnja A, Milenovic N, Lukac S, Knezevic A, Klasnja J, Karan Rakic V. The Effects of Regular Physical Activity and Playing Video Games on Reaction Time in Adolescents. Int J Environ Res Public Health. 2022 Jul 29;19(15):9278. doi: 10.3390/ijerph19159278. PMID 35954637